CLINICAL TRIAL: NCT00186433
Title: A Longitudinal Study of Plasma EBV DNA in Nasopharyngeal Carcinoma From Both Endemic and Non-Endemic Patient Populations
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Quynh-Thu Le, Katharine Dexter McCormick and Stanley McCormick Memorial Professor, Stanford University
Other Study IDs: ENT0006; ENT0006 (Other: Stanford University); 77622 (Other: Stanford University Alternate IRB Approval Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Mouth Cancer; Lip Cancer; Throat Cancer; Lip Neoplasms; Head and Neck Cancers
MeSH Terms: conditions — Mouth Neoplasms; Lip Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. To determine the prognostic implication of plasma Epstein-Bar Virus (EBV) DNA concentrations, as measured by quantitative polymerase chain reaction (PCR) in patients with nasopharyngeal carcinoma (NPC).
2. To relate pretreatment plasma EBV DNA concentration to WHO classification of these tumors both in endemic and non-endemic areas.
3. To determine whether pretreatment plasma EBV DNA can serve as a prognostic factor for both endemic and non-endemic patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Having a new diagnosis of Nasopharyngeal carcinoma.
* Being treated with either radiotherapy or chemoradiotherapy for this condition.

Exclusion Criteria:

* Age <18 since NPC is a very rare condition in this age group and may have a different biological behavior
* Patients who are unable to provide informed consents for themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Having a new diagnosis of Nasopharyngeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2001-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Plasma Epstein-Bar Virus (EBV) DNA concentrations | every 6 months until end of study
  measured by quantitative polymerase chain reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Le QT, Zhang Q, Cao H, Cheng AJ, Pinsky BA, Hong RL, Chang JT, Wang CW, Tsao KC, Lo YD, Lee N, Ang KK, Chan AT, Chan KC. An international collaboration to harmonize the quantitative plasma Epstein-Barr virus DNA assay for future biomarker-guided trials in nasopharyngeal carcinoma. Clin Cancer Res. 2013 Apr 15;19(8):2208-15. doi: 10.1158/1078-0432.CCR-12-3702. Epub 2013 Mar 4. PMID 23459720